CLINICAL TRIAL: NCT06620640
Title: A Randomized, Double-blind, Experimental Study Evaluating the Efficiency and Safety for the VGuard Device in the Treatment of Alzheimer's Disease.
Brief Title: A Study Evaluating the Efficiency and Safety for the VGuard Device in Alzheimer's Disease.
Acronym: CogniGuard
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuromedical Sp. z o.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VGuard- MCI- AD- 2020
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Alzheimer Disease (AD)
Keywords: Alzheimer Disease (AD)
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A: Active VGuard device (Experimental): Active VGuard device
  Interventions: Device: Intervention will most probably modify activity of neuron networks in specific brain areas responsible for cognitive functions, especially memory consolidation.
- ARM B: Sham VGuard device (Sham Comparator): Sham VGuard device
  Interventions: Device: Intervention will most probably modify activity of neuron networks in specific brain areas responsible for cognitive functions, especially memory consolidation.

INTERVENTIONS:
Device: Intervention will most probably modify activity of neuron networks in specific brain areas responsible for cognitive functions, especially memory consolidation. — Nigth stimulation

SUMMARY:
The project will allow the assessment of the safety and clinical effectiveness of the device for the treatment of cognitive impairment at Alzheimer's diease. The technology used in this study is based on the vagal nerve stimulation method used for more than 25 years and approved by the FDA in the treatment of drug-resistant epilepsy, depression and migraine. The study will use a non-invasive device for percutaneous electrostimulation of the vagal nerve. The previous clinical experience described in the literature has shown that vagal nerve stimulation leads to the activation of brain areas responsible for processing and consolidation of the fresh memory, i.e. the memory being impaired in so-called Alzheimer's Disease -AD. In relation to currently used methods of cognitive disorders treatment such as pharmacotherapy, the new solution will increase the effectiveness of therapy. In addition, VGuard is a completely non-invasive device that uses percutaneous stimulation, safe for the patient, and stimulation ranges are below the threshold of perception.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent prior to beginning study-related procedures.
2. Female and male subjects aged ≥ 60
3. Able to comply with the study protocol, in the investigator's judgment.

Exlusion Criteria:

1. Current or past history of: active psychosis, intellectual disability, bipolar disorder, alcohol abuse, addiction to psychoactive substances or any other major psychiatric condition.
2. Current or past history of any neurological disorder other than dementia, such as: epilepsy, stroke, Transient Ischemic Attack (TIA), Huntington's disease, Hakim syndrome, Parkinson's disease, multiple sclerosis, intracranial hematoma or brain lesions; and history of previous neurosurgery or head trauma that resulted in residual neurologic impairment.
3. Anticancer treatment within 12 months prior to the screening visit.
4. Clinically relevant serious co-morbid medical conditions within 3 months prior to the screening visit, including, but not limited to:

   1. current active or persistent infection
   2. clinically significant cardiac disease including unstable angina, acute myocardial infarction, congestive heart failure (NYHA III or NYHA IV), uncontrolled arrhythmia, uncontrolled hypertension (> 2nd stage),
   3. severe liver disease
   4. severe renal impairment
   5. uncontrolled diabetes
   6. chronic obstructive pulmonary disease (COPD)
   7. other metabolic, endocrine or systemic diseases affecting the central nervous system (present hypothyroidism), which in the physician's opinion may be the cause of dementia.
5. Permanent usage of benzodiazepines or cholinergic drugs.
6. Insomnia
7. Metal implants (excluding dental fillings) or devices such as pacemaker, medication pump, nerve stimulator, TENS unit, ventriculo-peritoneal shunt, cochlear implant, unless cleared by the study MD.
8. A serious communication barrier.
9. Clinically significant abnormalities at screening (Visit A) in laboratory tests, including: vitamin B12 deficiency or other laboratory abnormalities of possible clinical significance should be discussed with Principal Investigator to determine eligibility.

I 0. Positive pregnancy test ( for female of childbearing potential confirmed in medical interview) or is known from medical interview that woman is lactacting or pregnant.

11. Currently in a study of similar investigational device or investigational product which could interfere in study integrity.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Primary efficacy: proportion of patients responding to treatment with VGuard | up to 24 weeks
  The primary efficacy endpoint is defined as the proportion of patients responding to treatment with VGuard as measured by using the median change in the:
  * Mini-Mental State Examination (MMSE)
  * ADAS-cog
  scores from baseline between study arms. A responder is defined as a patient showing improvement or no decline in MMSE score on or from Visit C or E/F/G*.
  *Visit F and G will be performed according to Investigator's discretion.

SECONDARY OUTCOMES:
Secondary efficacy cognitive variable | up to 24 weeks
  The secondary efficacy endpoint is defined as the proportion of patients responding to treatment with VGuard as measured by using the median change in the:
  * Color Trails Test (CTT)
  * Verbal memory probing The scores from baseline between study arms. A responder is defined as a patient showing improvement or no decline in tests score from Visit C or E/F/G.* Responder rates will be evaluated separately for the listed above tests by independent raters.
    * Visit F will be performed according to Investigator's discretion.
Secondary efficacy affective and behavioral variables | up to 24 weeks
  Proportion of patients responding to treatment with VGuard between study arms.
  A responder is defined as a patient showing improvement or no decline in:
  * Hamilton Depression Rating Scale, HORS;
  * Satisfaction With Life Scale (SWLS) assessed at the following time-points:
  * VisitC
  * Visit D
  * Visit E + End of Study
  * Additional (Visit F/G*)
    * Visit F/G will be performed according to Investigator's discretion.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Adult Psychiatry Medical University of Lodz, Lodz, Łódź Voivodeship, Poland